CLINICAL TRIAL: NCT00952354
Title: Oral Language in Children With Down Syndrome: Lexical, Syntactic and Semantic Aspects
Brief Title: Oral Language in Children With Down Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Suelly Cecilia Olivan Limongi, University of São Paulo
Other Study IDs: 473492/2007-5; CNPq-473492/2007-5
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Down Syndrome
Keywords: Down syndrome; MLU; language development; language assessment
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- research group: 60 children aged from 3 to 10 years, both genders, observed in a symbolic play situation with their language therapists

SUMMARY:
The objective of this research is to verify the language of children with Down syndrome concerning lexical, syntactic and semantic aspects using MLU. The hypothesis is that children with Down syndrome will present low performance, regarding not only the quantitative measures as MLU-m, MLU-w, GM-1 and GM-2, but also regarding the qualitative aspects of their production, when compared to children with typical development.

DETAILED DESCRIPTION:
One of the alternatives to observe and assess language development and language disorders is to analyze spontaneous language samples, which allos the identification of qualitative and quantitative aspects. The analysis involves the MLU-morphemes, MLU-words and words classes. All words produced are analyzed, including interjections, adverbs and adjectives.Word classes with grammatical characteristics present lower averages, as prepositions and conjunctions. Reference parameters are the ones of the spoken language. The objective assessment with qualitative and quantitative data may help the speech and language pathologist/therapist to determine therapeutic guidelines to each patient.

ELIGIBILITY:
Inclusion Criteria:

* genetic diagnosis of Down syndrome
* good health conditions
* normal results on audiologic evaluation
* pediatric and ear, nose and throat periodic check ups.
* attend speech-language therapy at the Speech Language Pathology Laboratory in Syndromes and Sensorimotor Deficits (SLPL-SSD) of the School of Medicine of the University of São Paulo.

Exclusion Criteria:

* submission to long term hospitalizations due to heart diseases and major respiratory airway infections, that may interfere in the child's global development
* presence of visual or auditory important deficits

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 60 children with Down syndrome aged from 3 to 10 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Suelly CO Limongi, PhD, Study Chair — University of Sao Paulo; Rosangela V Andrade, PhD, Principal Investigator — University of Sao Paulo; Fabiola C Flabiano, PhD student, Principal Investigator — University of Sao Paulo; Porto Eliza, Ms student, Principal Investigator — University of Sao Paulo; Angela MA Carvalho, Ms student, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo - School of Medicine - Department of Physiotherapy, Communication Sciences and Disorders, Occupational Therapy, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Limongi SC, Oliveira Ede F, Ienne LM, Andrade RV, Carvalho AM. The use of nouns and verbs by children with Down syndrome in two different situations. Codas. 2013;25(3):262-7. doi: 10.1590/s2317-17822013000300012. English, Portuguese. PMID 24408338
- [Derived] Marques SF, Limongi SC. [Mean length utterance (MLU) as a measure of language development of children with Down syndrome]. J Soc Bras Fonoaudiol. 2011;23(2):152-7. doi: 10.1590/s2179-64912011000200012. Portuguese. PMID 21829931